CLINICAL TRIAL: NCT03670472
Title: Optimization of Correcting Molecules of Nonsense Mutations in Epithelial Cells of the Upper Airways of Patients With Cystic Fibrosis With Nonsense Mutations in the CFTR Gene
Brief Title: Correction of Nonsense Mutations in Cystic Fibrosis
Status: Recruiting | Type: Observational
Sponsor: University Hospital, Lille (Other)
Collaborators: Vaincre la Mucoviscidose (Other)
Responsible Party: Sponsor
Other Study IDs: 2013_59; 2014-A01236-41 (Other: ID-RCB number, ANSM)
Record Dates: First submitted 2018-08-01; First posted 2018-09-13 (Actual); Last update posted 2020-11-18 (Actual); Status verified 2020-10

CONDITIONS: Cystic Fibrosis
Keywords: Cystic fibrosis; nonsense mutations; CFTR gene; nasal epithelial cells; nonsense mutation readthrough
MeSH Terms: conditions — Cystic Fibrosis

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: smear of nasal fossae — 1 smear of nasal fossae during a usual or scheduled visit

SUMMARY:
The presence of a nonsense mutation leads to the rapid degradation of the carrier mRNA mutation by a mechanism called NMD (nonsense-mediated mRNA decay) [6, 13]. There are currently 3 main strategies at least for correcting nonsense mutations: exon skipping, inhibition of NMD and nonsense mutation readthrough.

In the laboratory, we developed a strategy for correcting nonsense mutations combining inhibition of NMD and activation of translecture. For this purpose, we have constructed screening systems to identify NMD-inhibiting and/or readthrough enhancers. The molecules thus identified are then tested on cell lines and in murine models carrying a nonsense mutation.

One of our goals is to select a set of molecules that can correct effectively nonsense mutations. For this we have to test these molecules on a great diversity of nonsense mutations.

This work will:

* determine if we can correct all the nonsense mutations tested with at least one of our molecules
* determine what is common within a group of mutations corrected by a given molecule
* be able to assign the parameters that make one mutation is corrected by one molecule and not or little by another.

This study will therefore improve our theoretical knowledge on the recognition of premature stop codons but also to propose therapeutic approaches for the correction of nonsense mutations of the CFTR gene in cystic fibrosis in a targeted way for a patient.

ELIGIBILITY:
Inclusion Criteria:

* Male / female adults and minors aged 8 years and over
* Patients with cystic fibrosis and carry a nonsense mutation on the 2 alleles of the gene coding for the CFTR channel.
* Patients whose genotype of patients concerning the CFTR gene is known.
* Patients with social security
* Major patients who have given their consent
* Minor patients with parental authorization

Exclusion Criteria:

* Patients who have a mutation other than nonsense in the CFTR gene
* Patients whose CFTR gene was not sequenced on the 2 alleles
* Patients not wishing to participate in this study or persons not giving or not able to give consent.
* Pregnant or lactating women
* Patients under curatorship or guardianship

Min Age: 8 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patients with cystic fibrosis and carry a nonsense mutation on the 2 alleles of the gene coding for the CFTR channel.
Sampling Method: Non-Probability Sample
Enrollment: 85 (Estimated)
Dates: Start 2016-02-03 (Actual); Primary Completion 2030-01 (Estimated); Study Completion 2030-01 (Estimated)

PRIMARY OUTCOMES:
Transport of iodide ions through the CEVAS membrane | less than 48hrs after the collect.
  Patient cells with be cultured in BEGM (Lonza) medium and incubated with corrector of nonsense mutations for 20 hours and with a fluorescent molecule called SPQ (for 6-methoxy-N-3'-sulfopropylquinolinium). Iodine can bind SPQ and will quench the SPQ fluorescence. Nitrates bind SPQ without quenching SPQ fluorescence. By placing patient cells first into an iodine-rich medium to quench the SPQ fluorescence and second into a nitrate-rich medium, we will be able to measure the level of functional CFTR protein present in these cells by measuring the re-apparition of fluorescence using fluorimeter. Indeed, nitrate will be able to replace iodine on SPQ without quenching SPQ fluorescence only if iodine exits cells through CFTR channels. This assay allows determining whether a corrector of nonsense mutation is able to lead to the synthesis of functional CFTR protein

SECONDARY OUTCOMES:
Immortalization of patient cells | an average 12 months
  Immortalization of patient cells will be attempted by transfection of construct expressing the origin-of-replication defective SV40 as described in Gruenert et al.,2004
Expression of the CFTR gene at the mRNA and protein level | less than 1 week.

CONTACTS AND LOCATIONS:
Overall Officials: Anne Prévotat, MD, Principal Investigator — University Hospital, Lille
Locations (8):
- France (8):
  - Camsp Chu Amiens, Amiens
  - Hopital Femme Mere Enfant - Hcl - Bron, Bron
  - Hôpital Calmette,CHU, Lille
  - Aphm Hopital La Timone - Marseille, Marseille
  - Chu Montpellier, Montpellier
  - Cmp Enfants Aphp Robert Debre - Paris, Paris
  - Hu Paris Centre Site Cochin Aphp - Paris 14, Paris
  - Hopitaux Universitaires de Strasbour, Strasbourg

IPD SHARING:
Plan to Share IPD: Undecided